CLINICAL TRIAL: NCT00231699
Title: A Comparison of Prevention of Hypothermia in Pediatric Patient Between Wrapping With Cotton (Webril) and Plastic (Mwrap).
Brief Title: A Comparison of Prevention of Hypothermia in Pediatric Patient Between Wrapping With Cotton and Plastic.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Prevention of Hypothermia
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2005-10-04 (Estimated); Status verified 2005-10

CONDITIONS: Perioperative Hypotension; Prevention; Child
Keywords: Prevention of Hypothermia; Pediatric Patient; Cotton; Plastic wrap
MeSH Terms: interventions — Control Groups

INTERVENTIONS:
Procedure: Plastic wrap (study group) and cotton (control group) wrap.

SUMMARY:
Hypothermia leads to increased morbidity and mortality. Heat loss mainly occurs during anesthesia and surgery. Therefore prevention of hypothermia in pediatric patients undergoing general anesthesia is very important. However, there is very little information about effectiveness of various insulating materials used in the operating room.

Objective: To compare the effectiveness of cotton and plastic for prevent intraoperative hypothermia in pediatric patients.

DETAILED DESCRIPTION:
A randomized controlled trial was conducted in 42 pediatric patients (age 1 month-3 years, ASA physical status 1-2) who were scheduled for elective maxillofacial or genitourinary surgery. The patients were randomly allocated into 2 groups. The patient's arms, legs and bodies were wrapped with either plastic (study group) or cotton (control group). All patients received standard general anesthesia with endotracheal tube and control ventilation with a fresh gas flow at 1 l/min. The core temperature (rectal temperature) was recorded every 10 minutes for 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 42 pediatric patients (age 1 month-3 years
* ASA physical status 1-2) who were scheduled for elective maxillofacial or genitourinary surgery.

Exclusion Criteria:

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42
Dates: Start 2004-01; Study Completion 2004-12

PRIMARY OUTCOMES:
Core temperature

CONTACTS AND LOCATIONS:
Overall Officials: waraporn chau-in, Asso Prof., Principal Investigator — Faculty of Medicine,KhonKaen University
Locations (1):
- Warporn Chau-in, KhonKaen, KhonKaen, Thailand